CLINICAL TRIAL: NCT06428123
Title: Comparison of Efficacy of Mirror Therapy vs Mental Imagery in Reduction of Phantom Limb Pain in Above Knee Amputee Patients: A Comparative Study
Brief Title: Comparison of Efficacy of Mirror Therapy vs Mental Imagery in Reduction of Phantom Limb Pain in AKAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/708
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Phantom Limb Pain
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror Therapy (Experimental)
  Interventions: Behavioral: Mirror Therapy on present Lower Limb
- Mental Imagery (Other)
  Interventions: Diagnostic Test: Mental Imagery on present Lower Limb

INTERVENTIONS:
Behavioral: Mirror Therapy on present Lower Limb — Patients will be seated close to a table on which a mirror will placed vertically. The normal (i.e., no amputated limb) will be placed in front of the mirror and made to perform movements of the different joints while the patient looking into the mirror.
  Arms: Mirror Therapy
Diagnostic Test: Mental Imagery on present Lower Limb — Mental imagery technique in which patients will be instructed to concentrate on sensations from each area of the body, including the phantom limb. Patients will be advised to imagine comfortable, thorough movement and sensation in the phantom limb, such that they could "stretch away the pain," and finally to "allow the limb to rest in a comfortable position." The actual therapy of "moving" and "feeling" the limb will lasted for 5 minutes. Patients will be asked to perform 40 minutes of meditation and imagery exercises.
  Arms: Mental Imagery

SUMMARY:
Limb amputation results in many types of pain, including localized pain at the stump and projected pain experienced by the patient in the location where the amputated limb used to be, known as phantom limb pain (PLP). The aim of this study is to determine the relative benefits of mirror therapy vs mental imagery in reduction of phantom limb pain. Randomized clinical trial study design will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female gender with ages from 12 to 75 years (17).
* Individuals with a unilateral above-knee amputation (AKA) at least 6 months prior to the study.
* Experiencing phantom limb pain at least 3 months (16).

Exclusion Criteria:

* History of neurological disorders affecting pain perception or motor function (e.g., stroke, spinal cord injury, brain injury).
* Uncontrolled diabetes or other medical conditions that could affect healing or participation in the study.
* Pregnancy or breastfeeding.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
The Numeric Rating (NRS) | 12 Months
  it is a simple and widely used tool for measuring pain intensity. It consists of a horizontal line with 11 numbered points, ranging from 0 (no pain) to 10 (worst pain imaginable). Patients are asked to rate their pain by selecting the number that best describes their current pain intensity

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Azra Naheed Medical College, Superior University, Lahore, Punjab Province
  - Ghurkee Hospital, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No